CLINICAL TRIAL: NCT03990233
Title: An Open-label Phase I Dose Finding Study of BI 765063, a Monoclonal Antibody (mAb) Antagonist of SIRPα, as Single Agent and in Combination With BI 754091, a Programmed Death-1 (PD-1) mAb, to Characterize Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy in Patients With Advanced Solid Tumours
Brief Title: A Trial of BI 765063 Monotherapy and in Combination With BI 754091 in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OSE Immunotherapeutics (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1443-0001; 2018-003830-34 (EudraCT Number)
Record Dates: First submitted 2019-05-21; First posted 2019-06-18 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor, Adult
Keywords: Checkpoint inhibitor (ICI); SIRPα; Advanced solid tumors; Anti-PD-1

STUDY DESIGN:
Intervention Model Description: * Step 1 (Dose escalation [Cohorts A and B]) primary objective : In V1/V1 homozygous and V1/V2 heterozygous patients with advanced solid tumors, Dose-Limiting Toxicities (DLTs), Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of BI 765063, as monotherapy (Cohort A) and in combination with BI 754091 (Cohort B).
  * Step 2 (Expansion Cohorts [Cohorts C]) primary objective : In V1/V1 homozygous patients with selected advanced solid tumors (colorectal or endometrium), DLT-like events and RP2D confirmation of BI 765063 in combination with BI 754091.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Step 1 (Dose escalation) : Cohorts A (Experimental): BI 765063 (SIRPα inhibitor) alone in V1/V1 homozygous and V1/V2 heterozygous patients with advanced solid tumours
  Interventions: Drug: BI 765063
- Step 1 (Dose escalation) : Cohorts B (Experimental): BI 765063 (SIRPα inhibitor) in combination with BI 754091 (PD-1 inhibitor) in V1/V1 homozygous and V1/V2 heterozygous patients with advanced solid tumours
  Interventions: Drug: BI 765063; Drug: BI 754091
- Step 2 (Expansion Cohorts) : Cohort C1 (Experimental): BI 765063 (SIRPα inhibitor) in combination with BI 754091 (PD-1 inhibitor) in V1/V1 homozygous patients with metastatic colorectal cancer
  Interventions: Drug: BI 765063; Drug: BI 754091
- Step 2 (Expansion Cohorts) : Cohort C2 (Experimental): BI 765063 (SIRPα inhibitor) in combination with BI 754091 (PD-1 inhibitor) in V1/V1 homozygous patients with metastatic endometrium cancer
  Interventions: Drug: BI 765063; Drug: BI 754091

INTERVENTIONS:
Drug: BI 765063 — mAb antagonist to SIRPα receptor, a myeloid checkpoint inhibitor
  Other Names: OSE-172
Drug: BI 754091 — mAb antagonist to PD-1 receptor, a lymphocyte T checkpoint inhibitor
  Arms: Step 1 (Dose escalation) : Cohorts B; Step 2 (Expansion Cohorts) : Cohort C1; Step 2 (Expansion Cohorts) : Cohort C2

SUMMARY:
This trial will be a two steps Phase I clinical study in patients with advanced solid tumors with an escalating phase (Step 1) followed by an expansion phase (Step 2) of BI 765063, a monoclonal antibody (mAb) antagonist to signal regulatory protein alpha (SIRPα) receptor, a myeloid checkpoint inhibitor administered as single agent, and in combination with BI 754091, a mAb antagonist to PD-1 receptor, a lymphocyte T checkpoint inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated, written informed consent form (ICF) prior to any trial-specific procedures.
2. Male or female aged ≥ 18 years (no upper limit of age) at the time of ICF signature.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy of at least 3 months.
5. Patients with a SIRPα polymorphism including at least one V1 allele will be selected (i.e., homozygous V1/V1 or heterozygous V1/V2 in separate cohorts in escalation [Step 1] and only homozygous V1/V1 in expansion cohorts [Step 2]); SIRPα polymorphism will be assessed in blood sampling (patient DNA) in a central laboratory; V1 allele is understood to include V1 and V1-like alleles.
6. In Step 1: Patients with histologically or cytologically documented advanced/metastatic primary or recurrent malignancies who failed or are not eligible to standard therapy;

   In Step 2: Cohort C1: Patients with histologically or cytologically advanced/metastatic primary or recurrent unresectable documented MSS colorectal tumors, whose disease relapsed after standard of care and who received no prior anti-PD-L1 inhibitors.

   Cohort C2: Patients with histologically or cytologically advanced or metastatic documented MSS endometrial carcinoma whose disease relapsed after standard of care and who received no prior anti-PD-L1 inhibitors.
7. Patients with at least one measurable lesion as per RECIST v1.1.
8. Patients must agree to pre- and on-treatment tumor biopsies. Fresh tumor biopsy may come either from the primary tumor or from a metastasis. Cytological material is not accepted. Archival tumor biopsy is acceptable, if done within 4 weeks before the first treatment administration.

   Biopsy sites should be carefully selected by the investigator so that it is safe for the patient and subsequent biopsy can be performed at the same location; also if possible should be distinct from the measurable lesion;
9. Adequate biological parameters defined as:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L.
   2. Hemoglobin (Hb) level ≥ 10 g/dL. (without recent red blood cell transfusion within 2 weeks prior to study entry)
   3. Platelet count ≥ 100 x 10^9/L.
   4. Total bilirubin level ≤ 1.5 X Upper Limit Normal (ULN), except for patients with Gilbert's syndrome from whom total bilirubin < 3.0 x ULN or direct bilirubin < 1.5 x ULN is authorized.
   5. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN.
   6. Serum creatinine ≤ 1.5 ULN; or creatinine clearance > 50 mL/min (Chronic Kidney Disease Epidemiology [CKD-EPI] formula).
   7. INR ≤ 1.5 (except if patient treated with anti-vitamin K); anticoagulation with anti-vitamin K and Low Molecular Weight Heparin [LMWH] is allowed;
10. Prior major treatment-related surgery completed at least 28 days before study drug administration;
11. In all cohorts :

    * An interval of at least 28 days since the last chemotherapy, approved immunotherapy, biological or investigational therapy, radiation or tyrosine kinase inhibitor (TKI) therapy (sunitinib, sorafenib) must have elapsed before the first study drug administration(s);
    * And all toxicities related to previous anticancer therapies have resolved to normal value or ≤ to Grade 1 prior to the study treatment administration, except alopecia.
12. Women must not be breastfeeding;
13. Women of childbearing potential (WOCB) must agree to use highly effective methods of contraception (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly), prior to study entry, during the study and for 5 months after the last dose of study drug.

    Highly effective methods of contraception are defined as one of the following methods: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomised partner, sexual abstinence.
14. Male patient with WOCBP partner must be willing to use male contraception (condoms) during the study and until 5 months after last dose of study drug. WOCBP partners of male subjects participating in the study may use hormone based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug (i.e.; oral hormonal contraception, cap, diaphragm, or sponge with spermicide).
15. Females of childbearing potential must have a serum negative pregnancy test within 7 days prior to first administration. Females who are postmenopausal for at least 1 year (defined as more than 12 months since last menses) or are surgically sterilized do not require this test.
16. Capable of understanding and complying with protocol requirements.
17. Patients must be affiliated to a social security system or an equivalent system.

Exclusion Criteria:

1. Patient with symptomatic/active central nervous system (CNS) metastases; Patient with previously treated brain metastases are eligible, if there is no evidence of progression for at least 28 days before the first study treatment administration, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period;
2. Other tumor location necessitating an urgent therapeutic intervention (e.g., palliative care, surgery or radiation therapy, such as spinal cord compression, other compressive mass, uncontrolled painful lesion, bone fracture).
3. Presence of other active invasive cancers, other than the one treated in this trial, within 5 years prior to screening.

   Except appropriately treated basal cell carcinoma of the skin, or in situ carcinoma of uterine cervix, or other local tumors considered cured by local treatment;
4. Patient with active autoimmune disease or a documented history of autoimmune disease, that requires systemic treatment (i.e. corticosteroids or immunosuppressive drugs).

   Except patients with vitiligo, resolved childhood asthma/atopy, alopecia, or any chronic skin condition that does not require systemic therapy, patients with autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone and/or controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
5. Known severe infusion related reactions to monoclonal antibodies (Grade ≥ 3 NCI-CTCAE v5.0) and patients removed from previous anti-PD-1 or anti-PD-L1 therapy because of a severe or life-threatening immune-related adverse event (irAE) (Grade ≥ 3 NCI-CTCAE v5.0);
6. Patients receiving systemic treatment with any immunosuppressive medication within one-week prior treatment start; Steroids of max. 10 mg prednisolone equivalent per day are allowed, topical and inhaled steroids are not considered as immunosuppressive.
7. Patients with interstitial lung disease or active, non-infectious pneumonitis.
8. Patient with uncontrolled disease-related metabolic disorders (e.g., hypercalcemia, SIADH) or uncontrolled diabetes;
9. Patient with uncontrolled congestive heart failure defined as New York Heart Association (NYHA) class III or IV, uncontrolled hypertension, unstable heart disease (e.g., coronary artery disease with unstable angina or myocardial infarction within 6 months before study treatment administration).
10. Patient with significant ECG abnormalities defined as any cardiac dysrhythmia (> Grade 2) (i.e., significant ventricular arrhythmia as persistent ventricular tachycardia and/or ventricular fibrillation; severe conduction disorders as atrio-ventricular block 2 and 3, sino-atrial block) or baseline QT/QTc interval >480 milliseconds (ms).
11. Patient with significant chronic liver disease (e.g., significant fibrosis, known cirrhosis) or active HBV or HCV infection; If HbsAg positive, an effective antiviral treatment to prevent hepatitis B reactivation is recommended.
12. Patients with known Human Immunodeficiency Virus (HIV) infection or patients with an active infection requiring specific anti-infective therapy until all signs of infection have resolved, and this within 2 weeks prior to the first study treatment administration;
13. Patient whose medical, psychological including alcohol or drug abuse, or surgical conditions are unstable and may affect the study completion and/or compliance and/or the ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Step 1 (dose escalation Parts A and B): Number of patients with Dose-Limiting Toxicities (DLTs) during the first treatment cycle | 3 weeks (1 cycle)
Step 1 (dose escalation Parts A and B): Maximum Tolerated Dose (MTD) determination | 3 weeks (1 cycle)
Step 2 (expansion combination Part C): Number of patients with DLT-like events during the whole treatment | An average of 1 year

SECONDARY OUTCOMES:
Step 1: Number of patients with DLT-like events during the whole treatment | An average of 1 year
Step 1 and 2: Incidence and severity of all Adverse Events (AEs), Serious AEs (SAEs), AEs of special interest (AESIs), Immune related AEs (irAEs) | An average of 1 year
Step 2: Objective Response Rate (ORR) defined as best response of Complete Response (CR) and Partial Response (PR) as per RECIST v 1.1 and immune RECIST (iRECIST) criteria | An average of 1 year
Step 1 and 2: Cmax determination | 12 weeks (4 cycles)
Step 1 and 2: AUC 0-tz determination | Up to 12 weeks (4 cycles)
Step 1 and 2: Percentage and evolution of SIRPα receptor occupancy (RO) in blood at pre, on-treatment and after the end of treatment | Up to 12 weeks (4 cycles)

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- France (5):
  - Institut Bergonie, Bordeaux
  - Hospital St Pierre, La Réunion
  - Centre Léon Berard, Lyon
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided